CLINICAL TRIAL: NCT02286583
Title: Early Detection of Breast Disease Using Medical Radiometer - RTM - 01 - RES
Brief Title: Medical Radiometer - RTM - 01 - RES and Its Use in Detecting Hotspots in Female Breast
Acronym: RTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Labdom Suisse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LabdomSuisseRD
Record Dates: First submitted 2014-10-18; First posted 2014-11-10 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: RTM; Female breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Microwave Thermography RTM-01-RES (No Intervention): Microwave thermography with sensitive probe that can detect skin and up to 8 cm microwave radiation deep tissues
  Interventions: Device: Microwave Thermography RTM-01-RES

INTERVENTIONS:
Device: Microwave Thermography RTM-01-RES — Divide the breast into 3 circles start from the nipple with 1 cm increase in the circle diameter. Divide this circle into 8 points. This makes us detect 24 points in addition to the nipple as fixed point and the tail of the breast as separate point giving total of 26 points.

SUMMARY:
Medical Radiometer depends on detecting the microwaves that radiates from deep structure hot objects in the body. When it comes to the breast, causes of deep structure hot spots are numerous, it can be inflammatory, hormonal or neoplastic. Therefore, the primary objective of this study is to test the sensitivity of the Medical Radiometer in detecting the hot spots in the breast.

DETAILED DESCRIPTION:
Several pathological lesions and physiological changes can cause spot in the breast to show higher temperature than it should be.

The causes can be:

[I] Physiological: During menarch, puberty, menstruation, lactation and after sexual Intercourse.

[II] Inflammatory: Mastitis and breast Abscess. [III] Endocrinal: any cause of increasing Oestrogen, Prolactin and/or Thyroid hormones.

[IV] Neoplastic: the neo-Vascularisation of the malignant tumors. Radiometer is a machine that can detect through its sensitive probe the microwave that radiate from the deep structures in the body.

The main aim of this study, first is to measure the sensitivity of the RTM in detecting the hot spots of different breast lesions.

The second Objective is to study the temperature patter of each disease trying to figure out a diagnostic code for the different lesions.

The tertiary objective is to combine the Echo-Dobbler in studying the hot spots in the neoplastic lesions trying to figure out an accurate protocol to early detect the malignant hot spots.

ELIGIBILITY:
Inclusion Criteria:

* The perfect sample should be 2000 females or more.
* 50 % already diagnosed breast cancer of any type
* 30% normal thought to be healthy females.
* 10% lactating
* 10% different breast diseases

Exclusion Criteria:

* Menstruating females.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Testing the sensitivity of the Microwave Thermography RTM-01-RES (ability to detect hotspots in breast lesions) | 6 months
  Ability of the Microwave Thermography RTM-01-RES to detect hotspots in the various breast lesions.

SECONDARY OUTCOMES:
Study the Temperature pattern | 3 months
  The temperature pattern of previously diagnosed diseases and the new healthy objects might give us an idea about whether we can diagnose various breast diseases or no.

OTHER OUTCOMES:
The detected hotspots, to be studdied by the Echo-dobbler to see the ability of early detection of neo-Vascularisation of the malignant tumors. | 6 months
  Half of the sample of the study will be already diagnosed cancer patients, study the neo-vascularisation of the tumor by the Echo-dobbler might give us an idea about how to detect the cancer in earlier stages when it is detected by the RTM

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alaa Abdelkarim M Mohammed Fouad, MRCGP [Int], Principal Investigator — Labdom Suisse
Locations (1):
- Poliklinik Permai Tanjumg Aru, Kota Kinabalu, Sabah, Malaysia